CLINICAL TRIAL: NCT03609944
Title: SpHincterotomy for Acute Recurrent Pancreatitis (SHARP Trial)
Brief Title: SpHincterotomy for Acute Recurrent Pancreatitis
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gregory Cote, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1922; U01DK116743 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pancreatitis; Pancreas Divisum; Pancreatitis, Acute; Pancreatitis Idiopathic; Pancreas Inflamed
Keywords: ERCP; Endoscopic retrograde cholangiopancreatography; pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreas Divisum | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to either EUS+sham or EUS+ERCP with miES.
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to the participant and the investigator assessing outcomes, study coordinators involved in collecting outcomes data will be masked to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS + Sham (Sham Comparator): Subjects randomized to EUS + sham will undergo a diagnostic endoscopic ultrasound (EUS) under sedation. The physician investigator will not make any attempts to achieve minor papilla cannulation, but photo document the minor papilla using a duodenoscope. Diluted dye will be injected into the duodenum. A small caliber prophylactic pancreatic duct stent will be deposited into the duodenal lumen. These maneuvers are performed to minimize the risk of unmasking.
  Interventions: Procedure: EUS
- EUS + ERCP with miES (Experimental): Subjects randomized to EUS + ERCP with miES will undergo the procedure at the same time as endoscopic ultrasound (EUS), under sedation. Indomethacin (100 mg) will be administered rectally at the onset of the ERCP procedure in patients with no known allergy to indomethacin. The techniques used to perform the endoscopic retrograde cholangiopancreatography (ERCP)with miES (minor papilla endoscopic sphincterotomy) will be left to the discretion of the study endoscopist. The extent of sphincterotomy will be per the discretion of the treating endoscopist. Unless methylene blue (or similar chromoendoscopy agent such as indigo carmine) has already been used to facilitate minor papilla cannulation, diluted dye will be injected into the duodenum.
  Interventions: Procedure: ERCP with miES; Procedure: EUS

INTERVENTIONS:
Procedure: ERCP with miES — Endoscopic retrograde cholangiopancreatography with minor papilla endoscopic sphincterotomy
  Arms: EUS + ERCP with miES
Procedure: EUS — Endoscopic ultrasound

SUMMARY:
The purpose of this study is to determine if a procedure called Endoscopic Retrograde CholangioPancreatography (ERCP) with sphincterotomy reduces the risk of pancreatitis or the number of recurrent pancreatitis episodes in patients with pancreas divisum. ERCP with sphincterotomy is a procedure where doctors used a combination of x-rays and an endoscope (a long flexible lighted tube) to find the opening of the duct where fluid drains out of the pancreas. People who have been diagnosed with pancreas divisum, have had at least two episodes of pancreatitis, and are candidates for the ERCP with sphincterotomy procedure may be eligible to participate. Participants will be will be randomly assigned to either have the ERCP with sphincterotomy procedure, or to have a "sham" procedure. Participants will have follow up visits 30 days after the procedure, 6 months after the procedure, and continuing every 6 months until a maximum follow-up period of 48 months.

DETAILED DESCRIPTION:
This is a sham-controlled, single blinded with a blinded outcome assessment, multi-center, randomized clinical trial of endoscopic retrograde cholangiopancreatography (ERCP) with minor papilla endoscopic sphincterotomy (miES) for the treatment of recurrent acute pancreatitis (RAP) with pancreas divisum. ERCP with miES is often offered in clinical practice to patients with RAP, pancreas divisum, and no other clear risk factors for their acute pancreatitis episodes. The hypothesis is that obstruction at the level of the minor papilla is one cause of RAP in pancreas divisum; miES will relieve the obstruction, thereby reducing the risk of a recurrent attack(s) of acute pancreatitis. The trial requires a total sample size of approximately 234 subjects, and a planned enrollment period of approximately 3.5 years with total planned study duration of 5 years (minimum follow-up of 6 months, maximum follow-up of 48 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must consent to be in the study and must have signed and dated an approved consent form.
2. >18 years
3. Two or more episodes of acute pancreatitis, with each episode meeting two of the following three criteria:

   * abdominal pain consistent with acute pancreatitis (acute onset of a persistent, severe, epigastric pain often radiating to the back)
   * serum lipase activity (or amylase activity) at least three times greater than the upper limit of normal
   * characteristic findings of acute pancreatitis on CECT, MRI or transabdominal ultrasonography
4. At least one episode of acute pancreatitis within 24 months of enrollment
5. Pancreas divisum confirmed by prior MRCP that is reviewed by an abdominal radiologist at the recruiting site.
6. By physician assessment, there is no certain explanation for recurrent acute pancreatitis.
7. Subjects must be able to fully understand and participate in all aspects of the study, including completion of questionnaires and telephone interviews, in the opinion of the clinical investigator

Exclusion Criteria:

1. Prior minor papilla therapy (endoscopic or surgical)
2. Calcific chronic pancreatitis, defined as parenchymal or ductal calcifications identified on computed tomography or magnetic resonance imaging scan that is reviewed by an expert radiologist at the recruiting site.
3. Main pancreatic duct stricture*
4. Presence of a structural etiology for acute pancreatitis, such as anomalous pancreatobiliary union, periampullary mass, or pancreatic mass lesion on imaging*
5. Presence of a local complication from acute pancreatitis which requires pancreatogram
6. Regular use of opioid medication for abdominal pain for the past three months
7. Medication as the etiology for acute pancreatitis by physician assessment
8. TWEAK score ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Cote, MD, MS, Study Chair — Oregon Health and Science University
Locations (21):
- United States (20):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Keck Hospital of USC, Los Angeles, California
  - Cedars-Sinai, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Luke's Hospital System, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of Rochester, Rochester, New York
  - The Ohio State University - Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Mason Hospital & Seattle Medical Center, Seattle, Washington
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cote GA, Durkalski-Mauldin VL, Serrano J, Klintworth E, Williams AW, Cruz-Monserrate Z, Arain M, Buxbaum JL, Conwell DL, Fogel EL, Freeman ML, Gardner TB, van Geenen E, Groce JR, Jonnalagadda SS, Keswani RN, Menon S, Moffatt DC, Papachristou GI, Ross A, Tarnasky PR, Wang AY, Wilcox CM, Hamilton F, Yadav D; SHARP Consortium. SpHincterotomy for Acute Recurrent Pancreatitis Randomized Trial: Rationale, Methodology, and Potential Implications. Pancreas. 2019 Sep;48(8):1061-1067. doi: 10.1097/MPA.0000000000001370. PMID 31404020
- [Background] Cote GA, Durkalski-Mauldin V, Williams A, Nitchie H, Serrano J, Yadav D; SHARP Consortium. Design and execution of sham-controlled endoscopic trials in acute pancreatitis: Lessons learned from the SHARP trial. Pancreatology. 2023 Mar;23(2):187-191. doi: 10.1016/j.pan.2022.12.011. Epub 2022 Dec 21. PMID 36585282
- [Derived] Cote GA, Durkalski-Mauldin V, Fogel EL, Moffatt DC, Wang AY, Lara LF, Tarnasky PR, Buxbaum JL, Dai SC, Jonnalagadda S, Willingham FF, Ross A, Keswani RN, Inamdar S, Kothari TH, Gardner TB, Jamidar PA, Gaddam S, Pleskow DK, Easler JJ, Elmunzer BJ, Coneys JG, Mallery JS, Strand DS, Papachristou GI, Slivka A, Kedia P, Sahakian AB, Kouanda A, Phan A, Williams A, Andersen DK, Serrano J, Yadav D; SHARP Consortium. Minor Papillotomy for Treatment of Idiopathic Acute Pancreatitis With Pancreas Divisum: A Randomized Clinical Trial. JAMA. 2026 Jan 14. doi: 10.1001/jama.2025.23988. Online ahead of print. PMID 41533371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EUS + Sham | EUS + ERCP With miES
Started | 73 | 75
Completed | 71 | 69
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EUS + Sham | EUS + ERCP With miES | Total
Number analyzed (Participants) | 73 | 75 | 148
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 52 [34 to 70] | 56 [35 to 77] | 54 [34.5 to 73.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 101
  Male | 21 | 26 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 66 | 71 | 137
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 65 | 64 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Reduce the Risk of Subsequent Acute Pancreatitis Episodes by 33%
Description: To test this aim, compare the incidence of acute pancreatitis > 30 days after treatment allocation as the primary outcome measure, using the next attack of acute pancreatitis as a time-to-event outcome.
Time Frame: This is a time-to-event outcome that is assessed starting 30 days after treatment through a maximum follow-up of 48 months.
Measure: Count of Participants; unit: Participants
Arm/Group | EUS + Sham | EUS + ERCP with miES
Number analyzed (Participants) | 73 | 75
Participants | 32 | 26

2. Secondary Outcome: To Compare the Incidence Rate Ratio of Acute Pancreatitis Between Treatment Groups
Description: All randomized subjects will be followed longitudinally until study completion (minimum follow-up of six months, maximum follow-up of 48 months), even if acute pancreatitis occurs during follow-up. A secondary benefit of miES may be a reduction in acute pancreatitis frequency, defined as the incidence rate (episodes/time pre- and post-randomization). Since baseline incidence rate is a probable predictor of post-randomization incidence rate, the investigators will compare the incidence rate ratios between the two arms, keeping person-time equal between the pre/post periods.
Time Frame: Incidence rate will be assessed starting 30 days after treatment through a maximum follow-up of 48 months.
Measure: Number (95% Confidence Interval); unit: Incidence rate ratio
Arm/Group | EUS + Sham | EUS + ERCP with miES
Number analyzed (Participants) | 73 | 75
Incidence rate ratio | 0.304 [.226 to .411] | .246 [.178 to .340]

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from randomization through the end of the 48-month study period. Non-serious adverse events were collected from randomization through Day 30.
Arm/Group | EUS + Sham | EUS + ERCP With miES
All-Cause Mortality (participants affected / at risk) | 3/73 | 2/75
Serious Adverse Events (participants affected / at risk) | 48/73 | 48/75
Other Adverse Events (participants affected / at risk) | 8/73 | 15/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUS + Sham (N=73) | EUS + ERCP With miES (N=75)
Missing (General disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 20 (59) | 25 (119)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 32 (82) | 31 (110)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (4)
Chest pain (General disorders and administration site conditions) | 0 (0) | 2 (2)
Death (General disorders and administration site conditions) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders and administration site conditions) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (5) | 3 (3)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Alcohol withdrawal syndrom (Psychiatric disorders) | 0 (0) | 1 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Pituitary tumour removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EUS + Sham (N=73) | EUS + ERCP With miES (N=75)
Missing (General disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders and administration site conditions) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT03609944/Prot_SAP_000.pdf